CLINICAL TRIAL: NCT03443531
Title: Effects of Traditional Chinese Medicine on Bronchiectasis Patients: A Multi-center, Randomized, Double-blind, Controlled Trial
Brief Title: Effects of Traditional Chinese Medicine on Bronchiectasis Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM for Bronchiectasis
Record Dates: First submitted 2018-01-26; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Traditional Chinese Medicine
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM (Experimental): Patients in this group will receive two types of TCM treatment, which are Bufei Huatan granule, Yifei Qinghua granule. The herbal extract twice daily for 24 weeks for lower dosage. The two granules are corresponding to the two traditional Chinese syndromes in sequence, which are syndrome of qi deficiency of lung and phlegm-turbidity obstructing the lung, Qi and Yin deficiency of the lung and the phlegm-heat obstructing the lung.
  Interventions: Drug: Bufei Huatan granule; Drug: Yifei Qinghua granule
- placebo TCM (Placebo Comparator): Patients in this group will be given two placebo TCM treatment, which are which are placebo Bufei Huatan granule, placebo Yifei Qinghua granule, corresponding to the two traditional Chinese syndromes in sequence, which are syndrome of qi deficiency of lung and phlegm-turbidity obstructing the lung, Qi and Yin deficiency of the lung and the phlegm-heat obstructing the lung.
  Interventions: Drug: Placebo Bufei Huatan granule; Drug: Placebo Yifei Qinghua granule

INTERVENTIONS:
Drug: Bufei Huatan granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of qi deficiency of lung and phlegm-turbidity obstructing the lung will be given Bufei Huatan granule, twice daily for 24 weeks for lower dosage.
  Arms: TCM
Drug: Yifei Qinghua granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of Qi and Yin deficiency of the lung and the phlegm-heat obstructing the lung will be given Yifei Qinghua granule, twice daily for 24 weeks for lower dosage.
  Arms: TCM
Drug: Placebo Bufei Huatan granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of qi deficiency of lung and phlegm-turbidity obstructing the lung will be given placebo Bufei Huatan granule, twice daily for 24 weeks for lower dosage.
  Arms: placebo TCM
Drug: Placebo Yifei Qinghua granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of Qi and Yin deficiency of the lung and the phlegm-heat obstructing the lung will be given placebo Yifei Qinghua granule, twice daily for 24 weeks for lower dosage.
  Arms: placebo TCM

SUMMARY:
The aim of this study is to evaluate the effectiveness of Traditional Chinese Medicine (TCM) on patients with clinically stable bronchiectasis by a multi-center, randomized, double-blind, controlled trial: one, TCM treatments based on syndrome differentiation; the other, a placebo of TCM treatment.

DETAILED DESCRIPTION:
Bronchiectasis is a common and frequently occurring respiratory disease, with more hospitalization rate and mortality, poor quality of life and heavy financial burden. The main clinical manifestations are persistent or recurrent cough, expectoration, sometimes accompanied by hemoptysis, which can cause respiratory dysfunction and chronic pulmonary heart disease. There are some randomized controlled trials of TCM for bronchiectasis, and have the effect in the treatment of bronchiectasis, reducing the number of acute aggravation and alleviating dyspnea. However, some TCM interventions lack comprehensive syndrome differentiation and the placebo control.

This is a multi-center, randomized, double-blind, controlled trial to compare the efficacy to evaluate the effectiveness of TCM on patients with clinically stable bronchiectasis. 216 subjects will be randomly assigned to one therapies (TCM treatments based on syndrome differentiation) and the other therapy (placebo of TCM treatment) for 24 weeks. After the treatment period, the subjects will be followed up for 24 weeks. The primary outcomes include the frequency of bronchiectasis exacerbation, and the secondary outcomes include quality of life (SGRQ, LCQ, QOL-B), pulmonary function, safety observation index.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of clinically stable bronchiectasis
* Age between 18 and 80 years
* Syndrome differentiation meets criteria of syndrome of Qi deficiency of lung and phlegm-turbidity obstructing the lung, syndrome of Qi and Yin deficiency of the lung and the phlegm-heat obstructing the lung
* Without participations in other interventional trials in the previous one month
* With the informed consent signed

Exclusion Criteria:

* Current respiratory disorders other than bronchiectasis (e.g. COPD,bronchial asthma, lung cancer,active tuberculosis, Interstitial lung disease, pulmonary thromboembolic, or Other patients who have an impact on the observation of disease)
* Patients with severe cardiovascular disease (e.g. Acute myocardial infarction,Acute heart failure)
* Severe liver disease(e.g.Active phase of hepatitis, Cirrhosis, Severe impairment of liver function by portal hypertension)
* Severe renal disease(e.g. renal transplant, dialysis)
* Patients with large hemoptysis in the last month
* Pregnant and lactating women
* Insanity, Dementia, and all kinds of Psychosis
* Smoking patients (Years of smoking10/ package year)
* Participating in other clinical trials with other interventions;
* Allergic to the used medicine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The frequency of bronchiectasis exacerbation | Changes in the frequency of exacerbation at the week 12 and week 24 of the treatment phase, and at the week 24 of the follow-up phase compared with baseline.
  The bronchiectasis exacerbations often result in reduced quality of life, increased rate of lung function decline, increased hospitalization. It is important to assess the changes of bronchiectasis exacerbations over time.

SECONDARY OUTCOMES:
The time to the first bronchiectasis exacerbation | Week 24 of the treatment phase.
Changes in Forced expiratory volume in one second | Changes in FEV1 at the week 24 of the treatment phase and the week 24 of the follow-up phase compared with baseline.
  Forced expiratory volume in one second (FEV1)is the amount of air that can be exhaled in one second. A positive change from baseline in FEV1 indicates improvement in lung function.

OTHER OUTCOMES:
Changes in St Georges respiratory questionnaire scores | Changes in the SGRQ scores at the week 12 and week 24 of the treatment phase, and the week 24 of the follow-up phase compared with baseline.
  Using the St Georges respiratory questionnaire (SGRQ) to asses the impact of Bronchiectasis on a person's life.
Changes in the Leicester Cough questionnaire scores | Changes in the LCQ scores at the week 12 and week 24 of the treatment phase, and the week 24 of the follow-up phase compared with baseline.
  Using the Leicester Cough questionnaire (LCQ) to asses the impact of Bronchiectasis on a person's life.
Changes in the Quality of Life-Bronchiectasis scores | Changes in the Qol-B scores at the week 12 and week 24 of the treatment phase, and the week 24 of the follow-up phase compared with baseline.
  Using the Quality of Life-Bronchiectasis (Qol-B) to asses the impact of Bronchiectasis on a person's life.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, Doctor, Study Chair — Henan University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No